CLINICAL TRIAL: NCT04196374
Title: Return of Genomic Results and Aggregate Penetrance in Population-Based Cohorts
Acronym: PopSeq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Framingham Heart Study (Unknown); Jackson Heart Study (Unknown); Broad Institute of MIT and Harvard (Other); University of Mississippi Medical Center (Other); Boston University (Other); Partners HealthCare (Other)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01HL143295 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Seemingly Healthy; Genetic Predisposition to Disease
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Intervention Model Description: Individuals who have had their DNA sequenced as part of TOPMed and are living will be notified if they have an actionable genomic result in an ACMG gene. There is no comparison group for this study.
Masking Description: There will be no masking all eligible individuals identified with an actionable genomic variant in an ACMG V2.0 gene will be notified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FHS & JHS participants with an actionable genomic finding (Experimental): Framingham and Jackson Heart Study participants who have had their genomes sequenced as part of TOPMed will be notified if an actionable genetic result in an ACMG v2.0 gene is identified and will be offered the opportunity to have their research result clinically confirmed by the study.
  Interventions: Genetic: Genomic Sequencing

INTERVENTIONS:
Genetic: Genomic Sequencing — Whole Genome Sequencing and reporting of actionable genomic results for genes included on the ACMG secondary findings list.

SUMMARY:
The PopSeq Project is a prospective cohort study that will develop and implement a genomic return of results (gRoR) process in the Framingham Heart Study (FHS) and Jackson Heart Study (JHS) cohorts and explore associated medical, behavioral, and economic outcomes. The study will interpret the genomic sequences of JHS/FHS participants previously sequenced by TOPMed who have consented to genomic return of results and/or genetic testing. We will develop and apply new methods for scalable screening/ classification of genomic variants and will explore genomic penetrance by phenotyping a subset of participants in the FHS and JHS.

DETAILED DESCRIPTION:
The objectives of this project are to: 1) Return clinically actionable genomic results to participants and track outcomes. Among living FHS/JHS participants who have consented to gRoR, we will contact those in whom a detrimental actionable variant is discovered in one of the genes noted on the ACMG recommended secondary findings list (estimate 2% of participants). 2) Improve high-throughput methods for identifying valid pathogenic variation. Refine and apply methods for high throughput screening of FHS/JHS genomes in a manner that retains high sensitivity for the detection of detrimental variants in ~3500 Mendelian disease-associated genes while reducing the false discovery rate of variants that are not pathogenic/likely pathogenic. 3) Explore aggregate penetrance for Mendelian diseases. Review phenotype data from a subset of FHS and JHS participants and compare this to genotypic data.

Data to be gathered include outcome and phenotypic data on the individuals who agree to gRoR and who learn that they have detrimental variant in one of the ACMG listed genes. These data will be self-reported through surveys and available medical records will be reviewed. Additional phenotypic data may be collected and reviewed for other non-actionable mendelian disease genes to explore genomic penetrance.

Research participants who are identified with a detrimental variant in an actionable gene may receive direct health benefits from learning this information; however, returning genomic results to healthy individuals not presenting for a medical indication may pose unexpected harms related to variant directed increases in screening and management. This study is focused on exploring the benefits and any potential harms related to returning genomic information in population-based cohorts. It will also allow us to better understand the penetrance of these variants in two populations not selected for disease status and will allow us to compare outcomes in a primarily African American population vs a Caucasian population. Developing methods to streamline variant analysis will help improve laboratory efficiency and will progress the field of variant curation and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Living individuals enrolled in the Framingham Heart Study and the Jackson Heart Study who have had their genomes sequenced as part of the TOPMed program.
* Adults over the age of 18 years
* Those who have consented to have their DNA samples used for research purposes (and those who participate in gRoR who have consented to receive genomic information).

Exclusion Criteria:

* Participants of the Framingham Heart Study or Jackson Heart Study who have not had their genomes sequenced as part of TOPMed
* Participants who did not opt for genomic/genetic research
* Participants who did/do not consent to receiving a genomic result (for the gRoR portion of this study only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Follow Through with Disclosure | From genetic result notification to 8 months post-disclosure
  JHS/FHS participants who have been sequenced through TOPMed, are alive and have consented for result return will be notified if an actionable genetic result is discovered. We will contact them and offer them the opportunity to have their research result clinically confirmed. We will evaluate the proportion of individuals who elect to have their result confirmed and disclosed to their health care provider.
Costs of Disclosure | 1 year post-disclosure
  We will determine the costs and associated time demands of implementing gRoR using a microcosting approach in which study staff track the amount of time they spend and the resources they use for each step of the protocol. For follow-up medical care, we will use a gross costing approach where we apply Centers for Medicare and Medicaid fee schedules to completed referrals and tests, hospitalizations and medication changes identified as described above.

SECONDARY OUTCOMES:
Guideline Compliance | History before disclosure
  Comparison of participants' personal and family histories of disease and their relevant available medical data against existing guidelines to identify instances where genetic testing and/or referral had been warranted but was never ordered.
New and Modified Diagnoses | 1 year post-disclosure
  We will examine cases to determine the percentage of individuals with a new or modified diagnosis attributed to results disclosure.
Self-Rated Health | Post disclosure and 1 year post-disclosure
  We will administer a single item of self rated health derived from the SF-12v2.
MD Recommendations | From disclosure to 1 month post-disclosure
  We will review chart notes from results disclosure sessions to determine services recommended in response to genetic findings.
Health Care Utilization | 1 year post-disclosure
  We will track health care utilization in response to results disclosure in the one year follow-up survey, including a) referrals and tests, b) hospitalizations, and c) medication changes

OTHER OUTCOMES:
Health Behaviors | 1 year post-disclsoure
  The survey includes a series of standardized yes/no questions to assess whether disclosed genetic information motivated participants to make changes to health behaviors. A summary score will be created based on the number of behaviors that participants report.
Disclosure-specific Impact | 6 months post-disclosure
  The survey assess the disclosure-specific impact of information on distress and positive emotions using an adapted 8-item version of the FaCTOR, a validated instrument developed for genomic sequencing that is sensitive to responses to high- and low-risk genetic risk results.
Satisfaction with Disclsoure | 6 months post-disclosure and 1 year post-disclosure
  Surveys will assess how helpful participants felt the results disclosure session was using a novel single question.
Decisional Regret | 6 months post-disclosure and 1 year post-disclosure
  Surveys will assess if participants regretted their decisions to receive their genetic findings using a novel single question.
Sharing with Relatives | 1 year post-disclsoure
  The survey will assess with how many relatives participants shared their genetic information.
Family Testing | 1 year post-disclsoure
  The survey will assess whether participants had relatives that received genetic testing based on disclosure to the participant.
General Anxiety | Post-disclosure and 6 months post-disclosure
  We will measure general anxiety using the General Anxiety Disorder Scale 2 (GAD-2), a validated 2-item instrument that will allow investigators to identify individuals with a potential mood disorder.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Framingham Heart Study, Framingham, Massachusetts
  - Jackson Heart Study, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Aggregate data will be shared through publication and will be considered upon request.

REFERENCES:
- [Background] Biesecker LG, Green RC. Diagnostic clinical genome and exome sequencing. N Engl J Med. 2014 Sep 18;371(12):1170. doi: 10.1056/NEJMc1408914. No abstract available. PMID 25229935
- [Background] Kalia SS, Adelman K, Bale SJ, Chung WK, Eng C, Evans JP, Herman GE, Hufnagel SB, Klein TE, Korf BR, McKelvey KD, Ormond KE, Richards CS, Vlangos CN, Watson M, Martin CL, Miller DT. Recommendations for reporting of secondary findings in clinical exome and genome sequencing, 2016 update (ACMG SF v2.0): a policy statement of the American College of Medical Genetics and Genomics. Genet Med. 2017 Feb;19(2):249-255. doi: 10.1038/gim.2016.190. Epub 2016 Nov 17. PMID 27854360
- [Background] Green RC, Berg JS, Grody WW, Kalia SS, Korf BR, Martin CL, McGuire AL, Nussbaum RL, O'Daniel JM, Ormond KE, Rehm HL, Watson MS, Williams MS, Biesecker LG; American College of Medical Genetics and Genomics. ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. Genet Med. 2013 Jul;15(7):565-74. doi: 10.1038/gim.2013.73. Epub 2013 Jun 20. PMID 23788249
- [Background] Wolf SM, Lawrenz FP, Nelson CA, Kahn JP, Cho MK, Clayton EW, Fletcher JG, Georgieff MK, Hammerschmidt D, Hudson K, Illes J, Kapur V, Keane MA, Koenig BA, Leroy BS, McFarland EG, Paradise J, Parker LS, Terry SF, Van Ness B, Wilfond BS. Managing incidental findings in human subjects research: analysis and recommendations. J Law Med Ethics. 2008 Summer;36(2):219-48, 211. doi: 10.1111/j.1748-720X.2008.00266.x. PMID 18547191
- [Background] Wolf SM, Crock BN, Van Ness B, Lawrenz F, Kahn JP, Beskow LM, Cho MK, Christman MF, Green RC, Hall R, Illes J, Keane M, Knoppers BM, Koenig BA, Kohane IS, Leroy B, Maschke KJ, McGeveran W, Ossorio P, Parker LS, Petersen GM, Richardson HS, Scott JA, Terry SF, Wilfond BS, Wolf WA. Managing incidental findings and research results in genomic research involving biobanks and archived data sets. Genet Med. 2012 Apr;14(4):361-84. doi: 10.1038/gim.2012.23. PMID 22436882
- [Background] Burke W, Evans BJ, Jarvik GP. Return of results: ethical and legal distinctions between research and clinical care. Am J Med Genet C Semin Med Genet. 2014 Mar;166C(1):105-11. doi: 10.1002/ajmg.c.31393. Epub 2014 Mar 10. PMID 24616381
- [Background] National Heart, Lung, and Blood Institute working group; Fabsitz RR, McGuire A, Sharp RR, Puggal M, Beskow LM, Biesecker LG, Bookman E, Burke W, Burchard EG, Church G, Clayton EW, Eckfeldt JH, Fernandez CV, Fisher R, Fullerton SM, Gabriel S, Gachupin F, James C, Jarvik GP, Kittles R, Leib JR, O'Donnell C, O'Rourke PP, Rodriguez LL, Schully SD, Shuldiner AR, Sze RK, Thakuria JV, Wolf SM, Burke GL. Ethical and practical guidelines for reporting genetic research results to study participants: updated guidelines from a National Heart, Lung, and Blood Institute working group. Circ Cardiovasc Genet. 2010 Dec;3(6):574-80. doi: 10.1161/CIRCGENETICS.110.958827. PMID 21156933
- [Background] Natarajan P, Gold NB, Bick AG, McLaughlin H, Kraft P, Rehm HL, Peloso GM, Wilson JG, Correa A, Seidman JG, Seidman CE, Kathiresan S, Green RC. Aggregate penetrance of genomic variants for actionable disorders in European and African Americans. Sci Transl Med. 2016 Nov 9;8(364):364ra151. doi: 10.1126/scitranslmed.aag2367. PMID 27831900
- [Background] Christensen KD, Phillips KA, Green RC, Dukhovny D. Cost Analyses of Genomic Sequencing: Lessons Learned from the MedSeq Project. Value Health. 2018 Sep;21(9):1054-1061. doi: 10.1016/j.jval.2018.06.013. Epub 2018 Aug 14. PMID 30224109
- [Background] Christensen KD, Vassy JL, Phillips KA, Blout CL, Azzariti DR, Lu CY, Robinson JO, Lee K, Douglas MP, Yeh JM, Machini K, Stout NK, Rehm HL, McGuire AL, Green RC, Dukhovny D; MedSeq Project. Short-term costs of integrating whole-genome sequencing into primary care and cardiology settings: a pilot randomized trial. Genet Med. 2018 Dec;20(12):1544-1553. doi: 10.1038/gim.2018.35. Epub 2018 Mar 22. PMID 29565423
- [Background] Roberts JS, Robinson JO, Diamond PM, Bharadwaj A, Christensen KD, Lee KB, Green RC, McGuire AL; MedSeq Project team. Patient understanding of, satisfaction with, and perceived utility of whole-genome sequencing: findings from the MedSeq Project. Genet Med. 2018 Sep;20(9):1069-1076. doi: 10.1038/gim.2017.223. Epub 2018 Jan 4. PMID 29300387
- [Background] Vassy JL, Christensen KD, Schonman EF, Blout CL, Robinson JO, Krier JB, Diamond PM, Lebo M, Machini K, Azzariti DR, Dukhovny D, Bates DW, MacRae CA, Murray MF, Rehm HL, McGuire AL, Green RC; MedSeq Project. The Impact of Whole-Genome Sequencing on the Primary Care and Outcomes of Healthy Adult Patients: A Pilot Randomized Trial. Ann Intern Med. 2017 Jun 27;167(3):159-169. doi: 10.7326/M17-0188. Print 2017 Aug 1. PMID 28654958
- [Background] Christensen KD, Dukhovny D, Siebert U, Green RC. Assessing the Costs and Cost-Effectiveness of Genomic Sequencing. J Pers Med. 2015 Dec 10;5(4):470-86. doi: 10.3390/jpm5040470. PMID 26690481
- [Background] Lupo PJ, Robinson JO, Diamond PM, Jamal L, Danysh HE, Blumenthal-Barby J, Lehmann LS, Vassy JL, Christensen KD, Green RC, McGuire AL; MedSeq Project team. Patients' perceived utility of whole-genome sequencing for their healthcare: findings from the MedSeq project. Per Med. 2016 Jan 1;13(1):13-20. doi: 10.2217/pme.15.45. Epub 2016 Jan 8. PMID 27019659
- [Background] Wolf SM, Branum R, Koenig BA, Petersen GM, Berry SA, Beskow LM, Daly MB, Fernandez CV, Green RC, LeRoy BS, Lindor NM, O'Rourke PP, Breitkopf CR, Rothstein MA, Van Ness B, Wilfond BS. Returning a Research Participant's Genomic Results to Relatives: Analysis and Recommendations. J Law Med Ethics. 2015 Fall;43(3):440-63. doi: 10.1111/jlme.12288. PMID 26479555
- [Background] McLaughlin HM, Ceyhan-Birsoy O, Christensen KD, Kohane IS, Krier J, Lane WJ, Lautenbach D, Lebo MS, Machini K, MacRae CA, Azzariti DR, Murray MF, Seidman CE, Vassy JL, Green RC, Rehm HL; MedSeq Project. A systematic approach to the reporting of medically relevant findings from whole genome sequencing. BMC Med Genet. 2014 Dec 14;15:134. doi: 10.1186/s12881-014-0134-1. PMID 25714468
- [Background] Machini K, Ceyhan-Birsoy O, Azzariti DR, Sharma H, Rossetti P, Mahanta L, Hutchinson L, McLaughlin H; MedSeq Project; Green RC, Lebo M, Rehm HL. Analyzing and Reanalyzing the Genome: Findings from the MedSeq Project. Am J Hum Genet. 2019 Jul 3;105(1):177-188. doi: 10.1016/j.ajhg.2019.05.017. Epub 2019 Jun 27. PMID 31256874
- [Background] Vassy JL, Lautenbach DM, McLaughlin HM, Kong SW, Christensen KD, Krier J, Kohane IS, Feuerman LZ, Blumenthal-Barby J, Roberts JS, Lehmann LS, Ho CY, Ubel PA, MacRae CA, Seidman CE, Murray MF, McGuire AL, Rehm HL, Green RC; MedSeq Project. The MedSeq Project: a randomized trial of integrating whole genome sequencing into clinical medicine. Trials. 2014 Mar 20;15:85. doi: 10.1186/1745-6215-15-85. PMID 24645908